CLINICAL TRIAL: NCT04154670
Title: An Open Label, Single Arm, Single Dose Study to Evaluate the Pharmacokinetics and Safety and Tolerability of MGTA 145 in Subjects With Normal Estimated GFR and Varying Degrees of Renal Impairment
Brief Title: Study Assessing PK and Safety of MGTA-145 in Subjects With Normal Estimated GFR and Varying Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ensoma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 145-RI-102
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Normal kidney function (Experimental): MGTA-145 single dose
  Interventions: Biological: MGTA-145
- Mild decrease in GFR (Experimental): MGTA-145 single dose
  Interventions: Biological: MGTA-145
- Moderate decrease in GFR (Experimental): MGTA-145 single dose
  Interventions: Biological: MGTA-145

INTERVENTIONS:
Biological: MGTA-145 — MGTA-145 will be given intravenously

SUMMARY:
This study is being conducted in healthy subjects and in subjects with a mild or moderate decrease in GFR (subjects with renal impairment).

DETAILED DESCRIPTION:
To investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of MGTA-145 in Subjects With Normal Estimated GFR and Varying Degrees of Renal Impairment

ELIGIBILITY:
Inclusion criteria for all subjects:

1. Age from 18 to 79 years, inclusive, at the time of signing of the ICF.
2. Body weight ≥50 kg and BMI 19 to 40 kg/m2, inclusive.
3. Systolic blood pressure ≤170 mmHg and diastolic blood pressure ≤100 mmHg at Screening and Day 1.
4. No clinically significant abnormalities on physical examination at Screening.
5. Alanine aminotransferase and aspartate aminotransferase up to 1.5 x the upper limit of normal (ULN) as long as total bilirubin and alkaline phosphatase are ≤ ULN.
6. No clinically significant abnormalities on ECG and QTcF <480 msec at Screening.
7. Female subjects are not pregnant, non-lactating, and must be of non-childbearing potential being either surgically sterile (eg, documented hysterectomy, bilateral oophorectomy, bilateral salpingo oopherectomy, tubal ligation) or post-menopausal women (over 45 years of age with 12 months or more amenorrhea verified by follicle stimulating hormone assessment and the absence of other biological or physiological causes).
8. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception (such as condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) after informed consent, throughout the study, and for a minimum of 90 days after the last dose, and who do not intend to donate sperm in the period from Screening until 3 months following administration of the study drug.
9. Subject using medications known to affect the elimination of serum creatinine (eg, cimetidine, trimethoprim) within the past 30 days.
10. Capable of providing informed consent and willing to comply with the requirements of the protocol.

    Specific inclusion criteria for subjects with NORMAL renal function:
11. Estimated GFR (based on MDRD equation) ≥90 mL/min/1.73 m2 (normal) as determined by an average of 2 values obtained at least 48 hours apart within the previous 3 months.
12. White blood cell (WBC) count, hemoglobin and platelet count within normal limits. Absolute neutrophil count of >1500/µL for African Americans and >2000/µL for other races.

    Specific inclusion criteria for subjects with RENAL IMPAIRMENT:
13. Estimated GFR <90 mL/min/1.73 m2 (based on MDRD equation) as determined by an average of 2 values obtained at least 48 hours apart and within the previous 3 months.
14. Stable renal function as determined by <20% difference in serum creatinine obtained on 2 occasions at least 48 hours apart and within the previous 3 months.
15. Platelet count ≥100,000/mm3, hemoglobin count ≥10g/dL, WBC count within normal limits. Absolute neutrophil count of >1500/µL for African Americans and >2000/µL for other races.

Exclusion criteria for all subjects:

1. Clinically significant abnormal finding on physical examination conducted at Screening. The assessment may be repeated once prior to treatment number assignment. If the repeat value(s) remains outside of protocol-specified ranges, the subject will be excluded from the study. Note: Re assessment is not allowed for subjects who have a positive urine drug screen test at Screening.
2. History of chronic alcohol or drug abuse within the previous 12 months. Subject has a positive pre-study drug/alcohol screen (to include at minimum: amphetamines, barbiturates, cocaine, opiates, cannabinoids, benzodiazepines, and myelosuppressive drugs). A subject with a positive finding on the drug screen may still be enrolled at the discretion of the Investigator if a plausible clinical explanation exists (eg, prior or concomitant medication use).
3. History of kidney transplantation or requiring dialysis or anticipated to initiate dialysis during the study period.
4. Donation of more than 500 mL of blood or plasma within 12 weeks prior to dosing.
5. Subject smokes more than 10 cigarettes per day (or equivalent) or has done so within 6 months prior to the Screening Visit.
6. Acute illness, infection (requiring medical treatment [eg, antibiotics]), or surgery within 30 days of dosing.
7. Seropositive for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus.
8. Subject has received another investigational drug or participated in an investigational device study within 30 days prior to dosing.
9. History of anaphylaxis or clinically important reaction to any drug including plerixafor.

   Specific exclusion criteria for subjects with NORMAL renal function:
10. Any clinically significant laboratory value outside the normal range at Screening. The assessment may be repeated once prior to treatment number assignment. If the repeat value(s) remains outside of protocol-specified ranges, the subject will be excluded from the study. Note: Re assessment is not allowed for subjects who have a positive urine drug screen test at Screening.
11. Any clinically significant hematologic, cardiovascular, pulmonary, central nervous system, metabolic, hepatic, or gastrointestinal conditions or history of conditions that, in the opinion of the Investigator may place the subject at an unacceptable risk as a participant in this study or may interfere with the interpretation of the study results.
12. Subject has used any prescription drugs within 14 days prior to dosing or any dietary supplements or non prescription drugs within 7 days prior to dosing unless deemed acceptable by the Investigator and Sponsor (Magenta Medical Monitor).

    Specific exclusion criteria for subjects with RENAL IMPAIRMENT:
13. Presence of acute kidney injury.
14. Clinically significant laboratory abnormalities excluding those associated with renal impairment or the underlying cause of renal disease.
15. Unstable medical condition or underlying medical condition that has changed within the past 90 days.
16. Presence of laboratory abnormalities or clinically significant medical condition that in the opinion of the Investigator may place the subject at an unacceptable risk as a participant in this study or may interfere with the interpretation of the study results.
17. Changes in prescription medications within 14 days prior to dosing or anticipated changes during the study period.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Biomarkers | 2 days
  Investigate area under the curve (AUC)
Pharmacokinetics Biomarkers | 2 days
  Investigate maximum plasma concentration (Cmax)
Pharmacokinetics Biomarkers | 2 days
  Investigate clearance (CL)
Pharmacokinetics Biomarkers | 2 days
  volume of distribution at steady state (Vdss)
Pharmacokinetics Biomarkers | 2 days
  Investigate half-life
Pharmacokinetics Biomarkers | 2 days
  Investigate renal clearance of MGTA-145

SECONDARY OUTCOMES:
Safety and Tolerability | 15 days
  Investigate the safety and tolerability of MGTA-145 following intravenous (IV) administration as monotherapy in subjects with varying degrees of renal impairment (e.g. adverse events, clinical laboratory tests, vital signs, ECGs)

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD, PhD, Study Director — Magenta Therapeutics
Locations (2):
- United States (2):
  - Orlando Clinical Research Center (OCRC), Orlando, Florida
  - Alliance for Multispeciality Research (AMR) Formerly New Orleans Center for Clinical Research (NOCCR), Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided